CLINICAL TRIAL: NCT03371342
Title: A Randomized, Double-blind, Active Controlled, Multi-center, Phase 1 Study to Investigate the Safety of MEDITOXIN® in Female Subjects With Idiopathic Overactive Bladder
Brief Title: Treatment of MEDITOXIN® in Female Patients With Idiopathic Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT01-KR17OAB101
Record Dates: First submitted 2017-11-28; First posted 2017-12-13 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDITOXIN (Experimental)
  Interventions: Drug: Meditoxin
- BOTOX (Active Comparator)
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Meditoxin — Meditoxin (Botulinum toxin type A)
  Arms: MEDITOXIN
Drug: Botox — Botox(Botulinum toxin type A)
  Arms: BOTOX

SUMMARY:
To investigate the safety of MEDITOXIN in female subjects with idiopathic overactive bladder compared with BOTOX

ELIGIBILITY:
Inclusion Criteria:

* Female aged more than 20 years
* Subject who has symptoms of Overactive Bladder for a period of at least 6 months immediately prior to screening

Exclusion Criteria:

- Patient not appropriate for participating in this study according to the investigator's opinion

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in adverse events of MEDITOXIN at 12 week | baseline, week 12 follow up visits
  safety profiles

SECONDARY OUTCOMES:
Change from baseline in the daily average number of episodes of urinary incontinence | baseline, week 12 follow up visits
  Urinary incontinence recorded by the participants in a bladder diary during the 3 consecutive days prior to the study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided